CLINICAL TRIAL: NCT00002033
Title: A Third-Party Blinded, Placebo Controlled Comparative Study of AS-101 Administered Intravenously in HIV Positive Patients With Advanced Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 045A; 753A-202-BR,MX
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-02

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; ammonium trichloro(dioxoethylene-O,O'-)tellurute; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; ammonium trichloro(dioxoethylene-O,O'-)tellurate

INTERVENTIONS:
Drug: Zidovudine
Drug: AS-101

SUMMARY:
To compare the effect of AS-101 to that of placebo on clinical efficacy and immunologic function in HIV positive patients with advanced disease. To compare the effect of AS-101 to that of placebo on occurrence of disease progression in HIV positive patients with advanced disease as defined by: (1) development of new diagnostically confirmed major opportunistic infection(s); or (2) development of AIDS-related dementia. To compare the effect of zidovudine (AZT) plus AS-101 versus AZT alone (placebo arm) on clinical efficacy and immunologic function in patients who require anti-viral therapy due to disease progression. Garlic capsules will be given to all study participants to mask the obvious garlic odor of AS-101.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Standard therapy including acyclovir or ganciclovir for infections that develop during the study period. (Prophylactic acyclovir is not permitted.) Standard therapy for persistent infections may continue.
* Immunomodulators or specific therapy for malignancies (including Kaposi's sarcoma) allowed only with permission of Wyeth-Ayerst medical monitor.
* Zidovudine (AZT) may be added only if there is disease progression and after the patient has been in the study for a minimum of eight weeks.
* Garlic capsules will be given to all study participants to mask side effects of AS-101.
* Required:
* Accepted standard prophylaxis for patients with prior Pneumocystis carinii pneumonia (PCP).

Patients must have the following:

* Diagnosis of AIDS or AIDS-related complex (ARC).
* Life expectancy > 6 months.
* Provide written informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Evidence of severe liver dysfunction (serum albumin < 2.5 g/dl, prothrombin time > 15 seconds or SGOT or SGPT > 3 x upper limits of normal), gastrointestinal, renal, respiratory, endocrine, hematologic, cardiovascular system abnormalities or psychiatric disorders which would prevent compliance with the protocol.
* Evidence of AIDS related dementia.
* Presence of disseminated Kaposi's sarcoma defined as any visceral lesions or > 20 cutaneous lesions; or Kaposi's sarcoma without at least one other AIDS defining characteristic.
* Presence of any lymphoma.
* Active opportunistic infection currently requiring treatment unless the infection has stabilized and continuing treatment is only required to prevent relapse (e.g., CNS toxoplasmosis or resolving tuberculosis).

Concurrent Medication:

Excluded:

* Prophylactic acyclovir.
* Immunomodulators or specific therapy for malignancies (including Kaposi's sarcoma) allowed only with permission of Wyeth-Ayerst medical monitor.
* Zidovudine (AZT) may be added only if there is disease progression and after the patient has been in the study for a minimum of eight weeks.

Patients with the following are excluded:

* Evidence of severe organ dysfunction as defined in Exclusion complications or other specified disease conditions.
* Unlikely or unable to comply with the requirements of the protocol.

Prior Medication:

Excluded within 8 weeks of study entry:

* Any immune stimulation agents such as BCG vaccine, interferons, or other immune modulators within 8 weeks.
* Any immunosuppressive agent within 8 weeks.
* Excluded within 12 weeks of study entry:
* Zidovudine (AZT).

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Escola Paulista De-Medicina, São Paulo
  - Faculdade De-Ciencias Medica Da, São Paulo
  - Hosp De-Servidor Publico Estadual, São Paulo
  - Instituto Do Cancer Arnaldo Vieiro, São Paulo

REFERENCES:
- [Background] Amarante JM, Levi GC, Pedro RJ, Galvao PA, Scheinberg M, Levy DS. A double blind controlled study with AS-101 in patients infected with HIV. Int Conf AIDS. 1992 Jul 19-24;8(2):B160 (abstract no PoB 3439)